CLINICAL TRIAL: NCT00133978
Title: REducing Deaths Due to OXidative Stress The REDOXS© Study
Brief Title: Trial of Glutamine and Antioxidant Supplementation in Critically Ill Patients
Acronym: REDOXS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daren K. Heyland (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Director, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REDOXS; EudraCT-No: 2007-001831-73
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Critical Illness; Sepsis; Multiple Organ Failure
Keywords: randomized trial; antioxidants; glutamine; organ failure
MeSH Terms: conditions — Critical Illness; Sepsis; Multiple Organ Failure | interventions — Glutamine; Antioxidants; alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Glutamine (Experimental): Glutamine supplementation
  Interventions: Other: Glutamine
- Antioxidants (Experimental): Antioxidant supplementation
  Interventions: Other: Antioxidants
- Glutamine + Antioxidants (Experimental): Glutamine and antioxidant supplementation
  Interventions: Other: Glutamine + Antioxidants
- Placebo (Placebo Comparator): Non-isonitrogenic, iso-caloric placebo solution
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Glutamine — 0.35 gm/kg/day parenterally and 30 gms/day enterally
  Arms: Glutamine
Other: Antioxidants — 500 micrograms of selenium/day parenterally and selenium 300 microgram, zinc 20 mg, beta carotene 10 mg, vitamine E 500 mg and vitamin C 1500 mg per day enterally
  Arms: Antioxidants
Other: Glutamine + Antioxidants — 0.35 g/kg/day glutamine parenterally and 30 g/day of glutamine enterally. 500 mcg selenium parenterally plus the following administered enterally: selenium 300 mcg, zing 20 mg, beta-carotene 10 mg, vitamin E 500 mg and vitamin C 1500mg
  Other Names: Dipeptiven, Microselenium/Selenium injection/selenase, EN REDOX formula (from Fresenius Kabi, Germany)
  Arms: Glutamine + Antioxidants
Other: Placebo — Normal saline intravenously and EN placebo formula (from Fresenius Kabi, Germany)
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether providing high dose glutamine and antioxidants to critically ill patients will be associated with improved survival.

DETAILED DESCRIPTION:
Background:

Critically ill patients experience a degree of hyperinflammation, cellular immune dysfunction, and oxidative stress. Supplementation with key nutrients, like glutamine and antioxidants, is most likely to have a favourable effect on these physiological parameters leading to an improvement in clinical outcomes. The results of two separate meta-analyses suggested that glutamine and antioxidants may be associated with improved survival. We have recently completed a dosing study to determine the maximal tolerable dose (MTD) of glutamine dipeptides and antioxidants in critically ill patients with evidence of hypoperfusion. The purpose of this protocol is to evaluate the effect of high dose glutamine and antioxidant supplementation on mortality in a large scale randomized trial.

Study Intervention:

Patients will be randomized to receive glutamine supplementation or antioxidant supplementation (or respective placebo).

ELIGIBILITY:
Inclusion Criteria:

* Mechanically ventilated patients > or = 18 years old
* 2 or more organ failures related to acute illness

Exclusion Criteria:

* > 24 hours from admission to ICU
* Patients who are moribund
* Lack of commitment to aggressive care
* Absolute contraindication to enteral nutrients
* Severe acquired brain injury
* Routine elective cardiac surgery
* Primary admission of burns > 30% body surface area
* Weight < 50 kgms or > 200 kgms
* Pregnant or lactating patients
* Previous randomization in this study
* Enrollment in a related ICU interventional study
* Child's class C liver disease
* Metastatic cancer with life expectancy < 6 months
* Seizure disorder requiring anticonvulsant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1223 (Actual)
Dates: Start 2005-04; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daren Heyland, MD, Study Chair — Clinical Evaluation Research Unit, Kingston General Hospital
Locations (34):
- United States (5):
  - Univ. of Colorado at Denver and Health Sciences Center, Aurora, Colorado
  - University of Louisville, Louisville, Kentucky
  - Miami Valley Hospital, Dayton, Ohio
  - University of Texas, Houston, Texas
  - Fletcher Allan Centre, Burlington, Vermont
- Belgium (2):
  - UZ Brussels, Brussels
  - University Hospital, Liège
- Canada (21):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Grey Nun's Hospital, Edmonton, Edmonton, Alberta
  - Vancouver Hospital, Vancouver, British Columbia
  - St Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Health Science Centre, Winnipeg, Manitoba
  - Capital Health Queen Elizabeth II HSC, Halifax, Nova Scotia
  - St Joseph's Healthcare, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London HSC Victoria Campus, ON, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Ottawa Hospital Civic Hospital, Ottawa, Ontario
  - Sunnybrook & Women's College, Toronto, Toronto, Ontario
  - Mt Sinai Hospital, Toronto, Ontario
  - Hopital Maisonneuve-Rosemount, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General, Montreal, Quebec
  - Hopital de Sacre-Coeur, Montreal, Quebec
  - Enfant-Jesus, Québec
- Germany (4):
  - Universitatsklinikum der Ernst-Moritz-Arndt-Universitat, Greifswald
  - Asklepios Kliniken Hamburg Altona, Hamburg
  - University Medical Center Schleswig-Holstein, Kiel
  - Universitatsklinikum Schleswig-Holstein Campus Luebeck, Lübeck
- Switzerland (2):
  - CHUV, Lausanne
  - University of Zurich, Zurich

REFERENCES:
- [Background] Heyland DK, Dhaliwal R, Drover JW, Gramlich L, Dodek P; Canadian Critical Care Clinical Practice Guidelines Committee. Canadian clinical practice guidelines for nutrition support in mechanically ventilated, critically ill adult patients. JPEN J Parenter Enteral Nutr. 2003 Sep-Oct;27(5):355-73. doi: 10.1177/0148607103027005355. PMID 12971736
- [Background] Heyland DK, Dhaliwal R, Suchner U, Berger MM. Antioxidant nutrients: a systematic review of trace elements and vitamins in the critically ill patient. Intensive Care Med. 2005 Mar;31(3):327-37. doi: 10.1007/s00134-004-2522-z. Epub 2004 Dec 17. PMID 15605227
- [Background] Novak F, Heyland DK, Avenell A, Drover JW, Su X. Glutamine supplementation in serious illness: a systematic review of the evidence. Crit Care Med. 2002 Sep;30(9):2022-9. doi: 10.1097/00003246-200209000-00011. PMID 12352035
- [Result] Heyland D, Muscedere J, Wischmeyer PE, Cook D, Jones G, Albert M, Elke G, Berger MM, Day AG; Canadian Critical Care Trials Group. A randomized trial of glutamine and antioxidants in critically ill patients. N Engl J Med. 2013 Apr 18;368(16):1489-97. doi: 10.1056/NEJMoa1212722. PMID 23594003
- [Derived] Heyland DK, Elke G, Cook D, Berger MM, Wischmeyer PE, Albert M, Muscedere J, Jones G, Day AG; Canadian Critical Care Trials Group. Glutamine and antioxidants in the critically ill patient: a post hoc analysis of a large-scale randomized trial. JPEN J Parenter Enteral Nutr. 2015 May;39(4):401-9. doi: 10.1177/0148607114529994. Epub 2014 May 5. PMID 24803474
- See also: Click here for more information about this study: A Randomized Trial of Glutamine and Antioxidant Supplementation in Critically Ill Patients — http://www.criticalcarenutrition.com/index.php?option=com_content&task=view&id=19&Itemid=42

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted between April 2005 and December 2011 in 40 ICUs in participating countries after local jurisdictional and institutional Research Ethics Board approval.
Pre-assignment Details: Written informed consent was obtained from patients or their legal representatives before enrollment.
Groups:
- Glutamine: Glutamine supplementation 0.35 g/kg/day of glutamine intravenously based on ideal body weight, provided as 0.50 g/kg/day of the dipeptide alanyl-glutamine and 30 g/day enterally, provided as alanyl-glutamine and glycine-glutamine dipeptides.
- Antioxidants: Antioxidant supplementation 500 ug of selenium intravenously, and the following vitamins and minerals enterally-- selenium 300 g, zinc 20 mg, beta carotene 10 mg, vitamin E 500 mg, and vitamin C 1500 mg.
- Glutamine + Antioxidants: Glutamine and antioxidant supplementation 0.35 g/kg/day of glutamine intravenously based on ideal body weight, provided as 0.50 g/kg/day of the dipeptide alanyl-glutamine and 30 g/day enterally, provided as alanyl-glutamine and glycine-glutamine dipeptides.
  500 ug of selenium intravenously , and the following vitamins and minerals enterally-- selenium 300 g, zinc 20 mg, beta carotene 10 mg, vitamin E 500 mg, and vitamin C 1500 mg.
Period: Overall Study
Arm/Group | Glutamine | Antioxidants | Glutamine + Antioxidants | Placebo
Started | 303 | 308 | 310 | 302
Completed | 301 | 307 | 310 | 300
Not Completed | 2 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Five randomized patients were not evaluable because we could not ascertain their 28-day vital status leaving 1218 patients in the final intention-to-treat analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Glutamine | Antioxidants | Glutamine + Antioxidants | Placebo | Total
Number analyzed (Participants) | 301 | 307 | 310 | 300 | 1218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 161 | 156 | 145 | 159 | 621
  >=65 years | 140 | 151 | 165 | 141 | 597
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (15.0) | 63.6 (14.3) | 64.3 (14.0) | 62.8 (13.7) | 63.3 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 130 | 130 | 122 | 492
  Male | 191 | 177 | 180 | 178 | 726
Region of Enrollment [Number; unit: participants]
  Canada | 259 | 262 | 263 | 260 | 1044
  United States | 32 | 34 | 34 | 31 | 131
  Germany | 6 | 6 | 5 | 4 | 21
  Belgium | 1 | 2 | 5 | 2 | 10
  Switzerland | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: 28-day Mortality
Description: 28-day mortality/status: at 28 days after randomization;
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | Glutamine | Antioxidants | Glutamine + Antioxidants | Placebo
Number analyzed (Participants) | 301 | 307 | 310 | 300
participants | 97 | 89 | 101 | 76

2. Secondary Outcome: ICU Length of Stay
Description: Measure of the duration of participant stay in the ICU
Time Frame: Day 28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Glutamine | Antioxidants | Glutamine + Antioxidants | Placebo
Number analyzed (Participants) | 301 | 307 | 310 | 300
days | 8.9 [5.6 to 16.0] | 8.9 [4.8 to 15.6] | 8.9 [5.0 to 15.1] | 8.3 [4.3 to 16.9]

3. Secondary Outcome: ICU Acquired Infection
Description: We have made some modifications the definitions developed by the International Sepsis Forum Consensus Conference (CCM 2005;33:1538-1548) to operationalize the adjudication of infections in this trial. We grade the certainty of the diagnosis of infection using definitions for 'Definite', 'Probable', and 'Possible' for each category of infection. The categories of infection are: Deep surgical wound infection, Incisional (or superficial) surgical wound infection, Skin and soft-tissue infection (non-surgical) (SSTS), Catheter-related blood stream infections (CRI), Primary blood stream infections (BSI), Lower urinary tract infection, Upper urinary tract infection, Intra abdominal infection, Sinusitis, Lower respiratory tract infection (excluding pneumonia), ICU Acquired Pneumonia and Other.
Time Frame: Day 28
Measure: Number; unit: participants
Groups:
- Glutamine: 0.35 g/kg/day of glutamine intravenously based on ideal body weight, provided as 0.50 g/kg/day of the dipeptide alanyl-glutamine and 30 g/day enterally, provided as alanyl-glutamine and glycine-glutamine dipeptides.
- No Glutamine; No Antioxidants: Non-isonitrogenic, iso-caloric placebo solution
- Antioxidants: 500 ug of selenium intravenously and the following vitamins and minerals enterally-- selenium 300 ug, zinc 20 mg, beta carotene 10 mg, vitamin E 500 mg, and vitamin C 1500 mg.
Arm/Group | Glutamine | No Glutamine | Antioxidants | No Antioxidants
Number analyzed (Participants) | 611 | 607 | 617 | 601
participants
  All Infections | 183 | 166 | 168 | 181
  Infections classified as 'definite' or 'probable' | 118 | 120 | 110 | 128
  Microbiological Confirmed | 92 | 87 | 83 | 96

4. Secondary Outcome: Hospital Length of Stay
Description: Measure of the duration of the participant's hospital stay
Time Frame: 6 months (from ICU admission)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Glutamine | Antioxidants | Glutamine + Antioxidants | Placebo
Number analyzed (Participants) | 301 | 307 | 310 | 300
days | 17.1 [9.0 to 35.1] | 16.0 [8.0 to 31.4] | 16.9 [8.2 to 37.0] | 16.5 [7.2 to 36.2]

ADVERSE EVENTS:
Time Frame: April 2005 and December 2011
Description: We collect data related to these hospitalized, critically ill patients' baseline illness in the CRF (e.g. abnormalities in oxygenation or ventilation, hemodynamic measures, etc). We reported changes in patients' baseline condition, events that are inconsistent with the underlying pathophysiology or progression of underlying disease, as SAEs.
Groups:
- Antioxidants: Antioxidant supplementation 500 ug of selenium intravenously and the following vitamins and minerals enterally-- selenium 300 ug, zinc 20 mg, beta carotene 10 mg, vitamin E 500 mg, and vitamin C 1500 mg.
- Glutamine + Antioxidants: Glutamine and antioxidant supplementation 0.35 g/kg/day of glutamine intravenously based on ideal body weight, provided as 0.50 g/kg/day of the dipeptide alanyl-glutamine and 30 g/day enterally, provided as alanyl-glutamine and glycine-glutamine dipeptides.
  500 ug of selenium intravenously and the following vitamins and minerals enterally-- selenium 300 ug, zinc 20 mg, beta carotene 10 mg, vitamin E 500 mg, and vitamin C 1500 mg.
Arm/Group | Glutamine | Antioxidants | Glutamine + Antioxidants | Placebo
Serious Adverse Events (participants affected / at risk) | 14/301 | 11/307 | 11/310 | 10/300
Other Adverse Events (participants affected / at risk) | 0/301 | 0/307 | 0/310 | 0/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Glutamine (N=301) | Antioxidants (N=307) | Glutamine + Antioxidants (N=310) | Placebo (N=300)
Nervous System Disorders (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2) | 2 (2)
Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Disorders (Cardiac disorders) | 7 (7) | 2 (2) | 5 (5) | 5 (5)
GI Disease (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3) | 5 (5)
Hepatobiliary Disorders (Hepatobiliary disorders) | 0 (0) | 0/301 (0) | 1 (1) | 0 (0)
Vascular Disorders (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye Disorders (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural Complications (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No